CLINICAL TRIAL: NCT04912856
Title: An Open-Label Extension of the Study XEN496 in Children With KCNQ2 Developmental and Epileptic Encephalopathy
Brief Title: An Open-Label Extension of the Study XEN496 (Ezogabine) in Children With KCNQ2-DEE
Acronym: EPIK-OLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision; not a safety decision
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPF-009-302; 2020-003447-28 (EudraCT Number)
Record Dates: First submitted 2021-05-03; First posted 2021-06-03 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Epilepsy; Epilepsy in Children; Epilepsy; Seizure; Disease; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Epileptic Syndromes
Keywords: XEN496; Ezogabine; Retigabine; Encephalopathy; Seizure; KCNQ2; EPIK
MeSH Terms: conditions — Epilepsy; Disease; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Epileptic Syndromes; Seizures | interventions — ezogabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will enter a blinded titration period (24 days) before moving to the open label treatment period for the remaining 35 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: XEN496 only (Experimental): 24-day blinded transition/titration period. Subjects who received XEN496 in the preceding study will continue to receive XEN496 at the same dose, in a blinded manner, without any further titration. To maintain the blinded aspect of the study, placebo will be dispensed to all subjects during the transition/titration period to ensure the total number of capsules are consistent across all subjects.
  Subjects who discontinue will be required to taper off study drug over a period of up to 15 days
  Interventions: Drug: XEN496
- Group 2: Placebo to XEN496 (Experimental): 24-day blinded transition/titration period. Subjects who were allocated to placebo in the preceding study, will be titrated to a tolerated dose up to a maximum dose of 21 mg/kg/day, with a maximum daily dose of 672 mg/day. To maintain the blinded aspect of the study, placebo will be dispensed to all subjects during the transition/titration period to ensure the total number of capsules are consistent across all subjects
  Subjects who discontinue or complete the study treatment will be required to taper off study drug over a period of up to 15 days.
  Interventions: Drug: XEN496

INTERVENTIONS:
Drug: XEN496 — XEN496 sprinkle capsules. Parents / caregivers will be instructed to sprinkle and mix the contents of the capsules into soft foods or liquids and feed it to the child.
  Other Names: ezogabine; retigabine

SUMMARY:
To assess the long-term safety and tolerability of XEN496 in pediatric subjects with KCNQ2 developmental and epileptic encephalopathy (KCNQ2-DEE) who had participated in the primary study (XPF-009-301).

DETAILED DESCRIPTION:
This is an open-label, long-term extension study of XEN496 for the treatment of seizures in subjects with KCNQ2-DEE, that will be open to eligible subjects who participated in the primary study, XPF-009-301. The primary objective is to assess the long-term safety of XEN496. A double-blind transition/titration period will be used to maintain blinding to the treatment allocation in the primary study (XPF-009-301). After completion of the blinded transition/titration period, subjects will receive the open label study drug at their optimal dose for approximately 35 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed participation in the primary study, XPF-009-301. A subject who withdraws from the primary study due to meeting protocol-specified worsening criteria will be considered as having completed participation in the primary study.
* The caregiver is willing and able to be compliant with diary completion, visit schedule, and study drug administration.
* Subject's caregiver achieved a minimum of 85% compliance with daily diary completion during both baseline and the double-blind period of the primary study.

Exclusion Criteria:

* Any adverse event(s) or serious adverse event(s) during the primary study XPF-009-301, which in the opinion of the investigator and sponsor's medical monitor, would preclude the subject's entry into the OLE study.
* A clinically significant condition or illness, or symptoms other than those resulting from KCNQ2-DEE, present at screening/baseline that, in the opinion of the investigator, would pose a risk to the subject if s/he were to enter the study.
* Any conditions that were specified as exclusion criteria in the primary study, XPF-009-301.
* It is anticipated that the subject will require treatment with at least 1 of the disallowed medications during the study.
* Any change in cardiac rhythm or atrioventricular conduction in the primary study that, in the investigator's opinion, is a significant risk to subject safety.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Xenon Pharmaceuticals Inc.
Locations (4):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - MultiCare Health System - Mary Bridge Pediatrics - Tacoma, Tacoma, Washington
- Sydney Children's Hospital, Sydney, New South Wales, Australia
- Universitair Ziekenhuis Antwerpen - Dienst Kinderneurologie, Edegem, Antwerpen, Belgium

REFERENCES:
- See also: XPF-009-301 Study (EPIK) — https://clinicaltrials.gov/ct2/show/NCT04639310

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: XEN496 Treatment in Preceding Study: 24-day blinded transition/titration period. Subjects who received XEN496 in the preceding study will continue to receive XEN496 at the same dose, in a blinded manner, without any further titration. To maintain the blinded aspect of the study, placebo will be dispensed to all subjects during the transition/titration period to ensure the total number of capsules are consistent across all subjects.
  Optimally-tolerated dose level established during the transition/titration period will be maintained throughout the duration of open-label period unless dose adjustment is required.
  Subjects who discontinue will be required to taper off study drug over a period of up to 15 days
  XEN496: XEN496 sprinkle capsules. Parents / caregivers will be instructed to sprinkle and mix the contents of the capsules into soft foods or liquids and feed it to the child.
  Placebo: Placebo sprinkle capsules. Parents / caregivers will be instructed to sprinkle and mix the contents of the capsules into soft foods or liquids and feed it to the child.
- Group 2: Placebo Treatment in Preceding Study: 24-day blinded transition/titration period. Subjects, who were allocated to placebo in the preceding study, will be titrated to a tolerated dose up to a maximum dose of 21 mg/kg/day, with a maximum daily dose of 672 mg/day. To maintain the blinded aspect of the study, placebo will be dispensed to all subjects during the transition/titration period to ensure the total number of capsules are consistent across all subjects.
  Optimally-tolerated dose level established during the transition/titration period will be maintained throughout the duration of open-label period unless dose adjustment is required.
  Subjects who discontinue will be required to taper off study drug over a period of up to 15 days
  XEN496: XEN496 sprinkle capsules. Parents / caregivers will be instructed to sprinkle and mix the contents of the capsules into soft foods or liquids and feed it to the child.
  Placebo: Placebo sprinkle capsules. Parents / caregivers will be instructed to sprinkle and mix the contents of the capsules into soft foods or liquids and feed it to the child.
Period: Overall Study
Arm/Group | Group 1: XEN496 Treatment in Preceding Study | Group 2: Placebo Treatment in Preceding Study
Started | 5 | 3
Completed | 1 | 0
Not Completed | 4 | 3
Not completed — Sponsor Decision; not due to safety reasons | 4 | 2
Not completed — Not reported in synoptic CSR. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: XEN496 Treatment in Preceding Study: 24-day blinded transition/titration period. Subjects who received XEN496 in the preceding study will continue to receive XEN496 at the same dose, in a blinded manner, without any further titration. To maintain the blinded aspect of the study, placebo will be dispensed to all subjects during the transition/titration period to ensure the total number of capsules are consistent across all subjects.
  Subjects who discontinue will be required to taper off study drug over a period of up to 15 days
  XEN496: XEN496 sprinkle capsules. Parents / caregivers will be instructed to sprinkle and mix the contents of the capsules into soft foods or liquids and feed it to the child.
- Group 2: Placebo Treatment in Preceding Study: 24-day blinded transition/titration period. Subjects, who were allocated to placebo in the preceding study, will be titrated to a tolerated dose up to a maximum dose of 21 mg/kg/day, with a maximum daily dose of 672 mg/day. To maintain the blinded aspect of the study, placebo will be dispensed to all subjects during the transition/titration period to ensure the total number of capsules are consistent across all subjects.
  Optimally-tolerated dose level established during the transition/titration period will be maintained throughout the duration of open-label period unless dose adjustment is required.
  Subjects who discontinue or complete the study treatment will be required to taper off study drug over a period of up to 15 days.
  XEN496: XEN496 sprinkle capsules. Parents / caregivers will be instructed to sprinkle and mix the contents of the capsules into soft foods or liquids and feed it to the child.
- Total: Total of all reporting groups
Arm/Group | Group 1: XEN496 Treatment in Preceding Study | Group 2: Placebo Treatment in Preceding Study | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 3 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 2 | 3
  United States | 3 | 1 | 4
  Australia | 1 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) Related to Intervention
Description: Safety and tolerability of XEN496 as assessed by incidence and severity of AEs and SAEs
Time Frame: From Screening/Baseline through to 4 weeks post last dose
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: XEN496 Treatment in Preceding Study | Group 2: Placebo Treatment in Preceding Study
Number analyzed (Participants) | 5 | 3
Participants
  Number of participants with any AEs | 5 | 3
  Number of participants with any TEAE | 5 | 3
  Participants with any treatment related TEAE | 1 | 2
  Participants with any TEAE leading to discontinuation of study drug | 0 | 0
  Participants with any TEAE leading to a dose reduction or treatment interruption | 1 | 1
  Participants with any Severe TEAE | 1 | 0
  Participants with any Serious TEAE | 2 | 1
  Participants with any TEAE leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: Collection of adverse event data began at Visit 1 when consent was obtained and continued throughout the course subject's participation in the study. The intended duration of the collection period was 3 years. Following the termination of the study, the collection period was up to 2 years and 3 months.
Arm/Group | Group 1: XEN496 Treatment in Preceding Study | Group 2: Placebo Treatment in Preceding Study
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/5 | 1/3
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: XEN496 Treatment in Preceding Study (N=5) | Group 2: Placebo Treatment in Preceding Study (N=3)
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Seizure cluster (Nervous system disorders) | 1 (2) | 0
Intestinal malrotation (Gastrointestinal disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: XEN496 Treatment in Preceding Study (N=5) | Group 2: Placebo Treatment in Preceding Study (N=3)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0
Alanine aminotransferase increased (Investigations) | 1 (1) | 0
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0
Retinal Pigmentation (Eye disorders) | 1 (1) | 0
Blood pressure systolic increased (Investigations) | 1 (1) | 0
Salivary gland enlargement (Gastrointestinal disorders) | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0
Swelling face (General disorders) | 1 (1) | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0
Pyrexia (General disorders) | 2 (2) | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0
Respiratory synctial virus test positive (Investigations) | 1 (1) | 0
Intestinal malrotation (Congenital, familial and genetic disorders) | 1 (1) | 0
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 (1) | 0
Blood in the stool (Gastrointestinal disorders) | 0 | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 | 1 (1)
Pneumonia (Infections and infestations) | 0 | 2 (3)
Urinary hesitation (Renal and urinary disorders) | 0 | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 | 2 (2)
Fatigue (General disorders) | 0 | 1 (1)
Initial Insomnia (Psychiatric disorders) | 0 | 1 (1)
Ear Swelling (Ear and labyrinth disorders) | 0 | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Bronchitis viral (Infections and infestations) | 0 | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 | 1 (1)
Epilepsy (Nervous system disorders) | 0 | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the early termination of the study (not due to safety reasons or futility) and the limited number of subjects enrolled in this OLE, the full analysis was not completed, and no efficacy data were assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT04912856/Prot_SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT04912856/SAP_002.pdf